CLINICAL TRIAL: NCT03322306
Title: Establishment of Genetic Basis for Neurological Disease by Genetic Screening and Development of Disease-specific Induced Pluripotent Stem (iPS) Cells From Dermal Fibroblasts in Selected Patients
Brief Title: Establishment of Genetic Basis for Neurological Disease by Genetic Screening
Status: Enrolling by invitation | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Anne YY CHAN, Associate Consultant, Chinese University of Hong Kong
Other Study IDs: iPS gene study CRE-2012.361
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Neuro-Degenerative Disease
Keywords: genetic screening; neuro-degenerative disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and skin sample will be saved for genetic test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Genechip screening kit — 10 ml blood for genetic screening by specific genetic screening kit

SUMMARY:
Hereditary neurological disorders are relatively common in paediatric neurological practice, but it has considerable overlap with adult neurological disorders. It is a group of of genetic diseases, most of which with a Mendelian inheritance affecting neurological system. Pathogenic mechanisms of these diseases are not fully understood. There is currently no effective therapy for most of these diseases. Disease-specific and patient- specific iPS cells would provide useful source of cells in culture modeling in these diseases.

In this study, disease-specific iPS cell lines repositories from hereditary neurological disease patients will be established. The cell lines will be registered and make them available to other investigators.

DETAILED DESCRIPTION:
The human iPS is generated by direct reprogramming of human somatic cells. These hiPS cells can give rise to most tissue types in the human embryo and possess many of the properties of human embryonic stem cells (hESC). The big advantage of human iPS cell over hESC is that it circumvents most of the limitations of hESC and remains the pluripotency for regeneration of cells and tissues. The unique capacity of self-renewal of iPS can provide unlimited supply of pluripotent stem cells for study. The patient-specific iPS cell lines should fundamentally eliminate the concern of immune rejection and ethical issues. The disease-specific iPS will facilitate the study of the mechanism of nucleotide expansion. It is the ideal medium to study the dynamic changes of the expansion from stem cell stage to different differentiation stages. It also creates a platform for drug development. The establishment of iPS stem cells will also make it realistic for target gene replacement/correction therapy.

Study subjects will be identified at the members from the Hong Kong Spinocerebellar ataxias (SCA) association and neurology clinic in Prince of Wales Hospital. Patients identify based on the diagnosis, genetic test results and inclusion and exclusion criteria.

10ml blood sample for genetic screening will be collected. Skin biopsy will only be scheduled if pathogenic mutation was identified by the genetic screening test and generation of iPS is considered necessary to study the pathogenic mechanism of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals at age 18 years or older who have presumed hereditary neurological disease.
2. Individuals or his/her guardian who can provide the informed consent.

Exclusion Criteria:

1. Individuals who are allergic to local anesthetics.
2. Individuals who have serious medical conditions that restrict their ability to tolerate skin biopsy.
3. Individuals who have history of bleeding diathesis or use of anticoagulant medications. Patients taking nonsteroidal anti-inflammatory agents will be asked to discontinue these medications 3 days prior to skin biopsy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have presumed hereditary neurological disease
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-11-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Specific genetic mutation | 1 year
  Able to identify disease-specific genetic mutation

CONTACTS AND LOCATIONS:
Overall Officials: Anne CHAN, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No